CLINICAL TRIAL: NCT00479388
Title: A Multicenter, Randomized, Double-Blind, Parallel Group, 12 Week Study to Evaluate the Efficacy and Safety of Extended-release (ER) Niacin/Laropiprant in Patients With Primary Hypercholesterolemia or Mixed Dyslipidemia.
Brief Title: Study of Extended Release Niacin/Laropiprant on Lipids (0524A-067)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0524A-067; 2007_521
Record Dates: First submitted 2007-05-24; First posted 2007-05-28 (Estimated); Results first posted 2009-07-31 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-02

CONDITIONS: Primary Hypercholesterolemia; Mixed Dyslipidemia
MeSH Terms: interventions — Simvastatin; Niacin; MK-0524; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Other): One tablet of ER niacin/ laropiprant (1g) + one tablet of the run-in statin dose, titrating up to ER niacin/laropiprant (2g) at Week 4 for an additional 8 weeks, with no adjustments to the run-in statin dose.
  Interventions: Drug: niacin (+) laropiprant
- 2 (Active Comparator): Stable dose of simvastatin or atorvastatin (20mg to 40mg) for 12 weeks.
  Interventions: Drug: Comparator: simvastatin; Drug: Comparator: atorvastatin calcium

INTERVENTIONS:
Drug: Comparator: simvastatin — simvastatin (20mg to 40mg) for 12 weeks.
  Other Names: Zocor®
  Arms: 2
Drug: niacin (+) laropiprant — One tablet of ER niacin/ laropiprant (1g); titrating up to ER niacin/laropiprant (2g) at Week 4 for an additional 8 weeks, with no adjustments to the run-in statin dose.
  Other Names: MK0524A
  Arms: 1
Drug: Comparator: atorvastatin calcium — atorvastatin calcium (20mg to 40mg) for 12 weeks.
  Other Names: atorvastatin
  Arms: 2

SUMMARY:
This is a 12-Week clinical trial in patients with Primary hypercholesterolemia or mixed dyslipidemia to study the effects of ER niacin/laropiprant on lipids.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 to 80 years of age with Primary hypercholesterolemia or mixed dyslipidemia
* Patients will be eligible for the study if their LDL-C values are within protocol specified range and meet other entry criteria

Exclusion Criteria:

* Patient whose LDL-C values are not within protocol specified range

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1216 (Actual)
Dates: Start 2007-07; Primary Completion 2008-07 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Shah S, Ceska R, Gil-Extremera B, Paolini JF, Giezek H, Vandormael K, Mao A, McCrary Sisk C, Maccubbin D. Efficacy and safety of extended-release niacin/laropiprant plus statin vs. doubling the dose of statin in patients with primary hypercholesterolaemia or mixed dyslipidaemia. Int J Clin Pract. 2010 May;64(6):727-38. doi: 10.1111/j.1742-1241.2010.02370.x. PMID 20518948
- [Derived] Bays HE, Shah A, Lin J, Sisk CM, Dong Q, Maccubbin D. Consistency of extended-release niacin/laropiprant effects on Lp(a), ApoB, non-HDL-C, Apo A1, and ApoB/ApoA1 ratio across patient subgroups. Am J Cardiovasc Drugs. 2012 Jun 1;12(3):197-206. doi: 10.2165/11631530-000000000-00000. PMID 22500948
- [Derived] Bays H, Shah A, Dong Q, McCrary Sisk C, Maccubbin D. Extended-release niacin/laropiprant lipid-altering consistency across patient subgroups. Int J Clin Pract. 2011 Apr;65(4):436-45. doi: 10.1111/j.1742-1241.2010.02620.x. PMID 21401833

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In: 30-Jul-2007 Last Patient Last Visit: 10-Jul-2008
  Investigators: 161 sites participated: Australia-5; Austria-4; Canada-11; Czech Republic-5; Denmark-4; France-10; Germany-24; Hungary-6; Israel-4; Italy-11; Netherlands-2; Norway-10; Poland-11; Russian Federation-7; South Africa-9; Spain-4; Sweden-17; United States-17
Pre-assignment Details: Patients on atorvastatin (10mg) or simvastatin (10mg or 20mg) had a 2 week run-in of their statin. Naïve patients or patients on other statins were started on simvastatin (10 or 20mg) or atorvastatin (10mg) for a 6 week run-in. Patients were eligible to be randomized if their Visit 1 low density lipoprotein cholesterol values were above goal.
Groups:
- ER Niacin/Laropiprant + Run-in Statin: One tablet of ER niacin/ laropiprant (1g) + one tablet of the run-in statin dose, titrating up to ER niacin/laropiprant (2g) at Week 4 for an additional 8 weeks, with no adjustments to the run-in statin dose.
- Run-in Statin Dose Doubled: Stable dose of simvastatin or atorvastatin (20mg to 40mg) for 12 weeks.
Period: Overall Study
Arm/Group | ER Niacin/Laropiprant + Run-in Statin | Run-in Statin Dose Doubled
Started | 606 | 610
Completed | 474 | 537
Not Completed | 132 | 73
Not completed — Adverse Event | 90 | 45
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Violation | 10 | 9
Not completed — Withdrawal by Subject | 32 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ER Niacin/Laropiprant + Run-in Statin | Run-in Statin Dose Doubled | Total
Number analyzed (Participants) | 606 | 610 | 1216
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (9.7) | 60.6 (9.8) | 60.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 304 | 289 | 593
  Male | 302 | 321 | 623
Coronary Heart Disease Risk Category by Goal [Number; unit: Participants]
  Low Risk at Goal | 27 | 26 | 53
  Low Risk Not at Goal | 16 | 14 | 30
  Multiple Risk at Goal | 91 | 82 | 173
  Multiple Risk Not at Goal | 92 | 71 | 163
  High Risk at Goal | 143 | 155 | 298
  High Risk Not at Goal | 237 | 262 | 499
Lipid Modification Type/Dose at Run-in [Number; unit: participants]
  Simvastatin 10 mg | 218 | 233 | 451
  Simvastatin 20 mg | 259 | 268 | 527
  Atorvastatin 10 mg | 129 | 109 | 238
Fasting Serum Glucose (FSG) [Mean (Standard Deviation); unit: mg/dL] | 108.3 (27.2) | 108.7 (27.7) | 108.5 (27.4)
High-density lipoprotein cholesterol [Mean (Standard Deviation); unit: mg/dL] | 54.89 (14.45) | 54.97 (13.91) | 54.93 (14.17)
Low-density lipoprotein cholesterol [Mean (Standard Deviation); unit: mg/dL] | 117.55 (28.66) | 115.82 (28.37) | 116.68 (28.52)
Triglycerides (TG) [Median (Full Range); unit: mg/dL] | 136.00 [46.00 to 594.00] | 124.00 [42.00 to 852.00] | 130.00 [42.00 to 852.00]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low Density Lipoprotein Cholesterol at Week 12
Time Frame: Baseline and 12 Weeks
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | ER Niacin/Laropiprant + Run-in Statin | Run-in Statin Dose Doubled
Number analyzed (Participants) | 572 | 595
Percent | -10.0 [-12.6 to -7.4] | -5.5 [-7.4 to -3.5]
Statistical Analysis 1: Comparison: ER Niacin/Laropiprant + Run-in Statin vs Run-in Statin Dose Doubled; Test type: Superiority or Other; p = 0.006, Repeated measures analysis; Study times: 4, 8 and 12 weeks. Terms: treatment-by-time, gender-by-time, baseline LDL-C-by-time and concomitant statin group-by-time interaction; Median Difference (Final Values) = -4.5, 95% CI [-7.7 to -1.3], Standard Error of Mean 1.6

2. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein Cholesterol at Week 12
Time Frame: Baseline and 12 Weeks
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | ER Niacin/Laropiprant + Run-in Statin | Run-in Statin Dose Doubled
Number analyzed (Participants) | 572 | 595
Percent | 15.8 [13.8 to 17.8] | 0.2 [-1.1 to 1.4]
Statistical Analysis 1: Comparison: ER Niacin/Laropiprant + Run-in Statin vs Run-in Statin Dose Doubled; Test type: Superiority or Other; p <= 0.001, Repeated measures analysis; Study times: 4, 8 and 12 weeks. Terms: treatment-by-time, gender-by-time, baseline HDL-C-by-time and concomitant statin group-by-time interaction; Mean Difference (Final Values) = 15.6, 95% CI [13.4 to 17.9], Standard Error of Mean 1.2

3. Secondary Outcome: Percent Change From Baseline in Triglycerides at Week 12
Time Frame: Baseline and 12 Weeks
Population: Full Analysis Set With at Least one Post-Titration Visit Measurement
Measure: Median (95% Confidence Interval); unit: Percent
Arm/Group | ER Niacin/Laropiprant + Run-in Statin | Run-in Statin Dose Doubled
Number analyzed (Participants) | 515 | 571
Percent | -17.6 [-21.0 to -14.2] | -4.0 [-7.2 to -0.9]
Statistical Analysis 1: Comparison: ER Niacin/Laropiprant + Run-in Statin vs Run-in Statin Dose Doubled; Test type: Superiority or Other; p <= 0.001, Repeated measures analysis; ANCOVA model based on Tukey's normalized ranks with term for treatment, gender, concomitant statin group and Tukey's normal score of baseline; Mean Difference (Final Values) = -15.4, 95% CI [-19.2 to -11.7]

ADVERSE EVENTS:
Arm/Group | ER Niacin/Laropiprant + Run-in Statin | Run-in Statin Dose Doubled
Serious Adverse Events (participants affected / at risk) | 14 | 8
Other Adverse Events (participants affected / at risk) | 249 | 172
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | ER Niacin/Laropiprant + Run-in Statin | Run-in Statin Dose Doubled
Acute coronary syndrome (Cardiac disorders) | 1/602 | 0/609
Acute myocardial infarction (Cardiac disorders) | 1/602 | 0/609
Cardiac failure congestive (Cardiac disorders) | 1/602 | 0/609
Eye discharge (Eye disorders) | 1/602 | 0/609
Chest pain (General disorders) | 0/602 | 1/609
Non-cardiac chest pain (General disorders) | 1/602 | 0/609
Drug hypersensitivity (Immune system disorders) | 1/602 | 0/609
Acute sinusitis (Infections and infestations) | 1/602 | 0/609
Oral herpes (Immune system disorders) | 1/602 | 0/609
Wound sepsis (Infections and infestations) | 1/602 | 0/609
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/602 | 1/609
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/602 | 0/609
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/602 | 1/609
Amnesia (Nervous system disorders) | 0/602 | 1/609
Cerebral haemorrhage (Nervous system disorders) | 0/602 | 1/609
Transient ischaemic attack (Nervous system disorders) | 0/602 | 1/609
Ovarian cyst (Reproductive system and breast disorders) | 1/602 | 0/609
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0/602 | 1/609
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0/602 | 1/609
Flushing (Vascular disorders) | 1/602 | 0/609
Hypotension (Vascular disorders) | 1/602 | 0/609
Peripheral ischaemia (Vascular disorders) | 1/602 | 0/609
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | ER Niacin/Laropiprant + Run-in Statin | Run-in Statin Dose Doubled
Anaemia (Blood and lymphatic system disorders) | 0/602 | 1/609
Neutropenia (Blood and lymphatic system disorders) | 0/602 | 2/609
Splenomegaly (Blood and lymphatic system disorders) | 0/602 | 1/609
Angina pectoris (Cardiac disorders) | 1/602 | 1/609
Arrhythmia (Cardiac disorders) | 0/602 | 1/609
Cardiac discomfort (Cardiac disorders) | 1/602 | 0/609
Palpitations (Cardiac disorders) | 1/602 | 2/609
Supraventricular extrasystoles (Cardiac disorders) | 1/602 | 0/609
Tachycardia (Cardiac disorders) | 0/602 | 1/609
Tinnitus (Ear and labyrinth disorders) | 0/602 | 1/609
Vertigo (Ear and labyrinth disorders) | 1/602 | 4/609
Cataract (Eye disorders) | 0/602 | 1/609
Conjunctivitis (Eye disorders) | 1/602 | 4/609
Dry eye (Eye disorders) | 1/602 | 0/609
Eye inflammation (Eye disorders) | 1/602 | 0/609
Eye irritation (Eye disorders) | 1/602 | 0/609
Eyelid oedema (Eye disorders) | 1/602 | 0/609
Lacrimation increased (Eye disorders) | 1/602 | 0/609
Retinal artery thrombosis (Eye disorders) | 0/602 | 1/609
Vision blurred (Eye disorders) | 0/602 | 1/609
Visual disturbance (Eye disorders) | 1/602 | 0/609
Abdominal distension (Gastrointestinal disorders) | 0/602 | 1/609
Abdominal pain (Gastrointestinal disorders) | 6/602 | 4/609
Abdominal pain lower (Gastrointestinal disorders) | 1/602 | 0/609
Abdominal pain upper (Gastrointestinal disorders) | 12/602 | 4/609
Anal fissure (Gastrointestinal disorders) | 0/602 | 2/609
Cheilitis (Gastrointestinal disorders) | 0/602 | 1/609
Constipation (Gastrointestinal disorders) | 1/602 | 6/609
Diarrhoea (Gastrointestinal disorders) | 16/602 | 4/609
Dry mouth (Gastrointestinal disorders) | 6/602 | 0/609
Duodenitis (Gastrointestinal disorders) | 2/602 | 0/609
Dyspepsia (Gastrointestinal disorders) | 7/602 | 5/609
Dysphagia (Gastrointestinal disorders) | 0/602 | 3/609
Eructation (Gastrointestinal disorders) | 1/602 | 0/609
Flatulence (Gastrointestinal disorders) | 1/602 | 3/609
Gastritis (Gastrointestinal disorders) | 2/602 | 1/609
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1/602 | 0/609
Haemorrhoids (Gastrointestinal disorders) | 0/602 | 2/609
Hiatus hernia (Gastrointestinal disorders) | 1/602 | 0/609
Hypoaesthesia oral (Gastrointestinal disorders) | 0/602 | 1/609
Nausea (Gastrointestinal disorders) | 20/602 | 9/609
Oral disorder (Gastrointestinal disorders) | 0/602 | 1/609
Stomach discomfort (Gastrointestinal disorders) | 1/602 | 0/609
Stomatitis (Gastrointestinal disorders) | 1/602 | 0/609
Toothache (Gastrointestinal disorders) | 2/602 | 0/609
Vomiting (Gastrointestinal disorders) | 7/602 | 4/609
Asthenia (General disorders) | 2/602 | 1/609
Chest discomfort (General disorders) | 0/602 | 1/609
Chest pain (General disorders) | 1/602 | 1/609
Chills (General disorders) | 1/602 | 1/609
Discomfort (General disorders) | 2/602 | 0/609
Fatigue (General disorders) | 1/602 | 2/609
Feeling cold (General disorders) | 0/602 | 1/609
Feeling hot (General disorders) | 9/602 | 3/609
Influenza like illness (General disorders) | 0/602 | 1/609
Malaise (General disorders) | 1/602 | 2/609
Non-cardiac chest pain (General disorders) | 1/602 | 1/609
Oedema peripheral (General disorders) | 2/602 | 3/609
Pain (General disorders) | 2/602 | 0/609
Pyrexia (General disorders) | 2/602 | 0/609
Cholelithiasis (Hepatobiliary disorders) | 0/602 | 1/609
Drug hypersensitivity (Immune system disorders) | 1/602 | 0/609
Acute tonsillitis (Infections and infestations) | 0/602 | 2/609
Balanitis candida (Infections and infestations) | 1/602 | 0/609
Breast abscess (Infections and infestations) | 0/602 | 1/609
Bronchitis (Infections and infestations) | 11/602 | 5/609
Bronchitis bacterial (Infections and infestations) | 0/602 | 1/609
Bronchopneumonia (Infections and infestations) | 1/602 | 1/609
Candidiasis (Infections and infestations) | 0/602 | 1/609
Cystitis (Infections and infestations) | 2/602 | 2/609
Ear infection (Infections and infestations) | 0/602 | 1/609
Furuncle (Infections and infestations) | 1/602 | 0/609
Gastroenteritis (Infections and infestations) | 3/602 | 6/609
Herpes simplex (Infections and infestations) | 1/602 | 0/609
Herpes zoster (Infections and infestations) | 2/602 | 1/609
Influenza (Infections and infestations) | 4/602 | 3/609
Mycoplasma infection (Infections and infestations) | 0/602 | 1/609
Nasopharyngitis (Infections and infestations) | 13/602 | 15/609
Oral herpes (Infections and infestations) | 1/602 | 0/609
Otitis media (Infections and infestations) | 2/602 | 0/609
Pharyngitis (Infections and infestations) | 1/602 | 0/609
Pulpitis dental (Infections and infestations) | 0/602 | 1/609
Respiratory tract infection (Infections and infestations) | 2/602 | 2/609
Rhinitis (Infections and infestations) | 1/602 | 0/609
Sinusitis (Infections and infestations) | 0/602 | 2/609
Tonsillitis (Infections and infestations) | 0/602 | 1/609
Tooth infection (Infections and infestations) | 0/602 | 1/609
Tracheobronchitis (Infections and infestations) | 1/602 | 2/609
Upper respiratory tract infection (Infections and infestations) | 5/602 | 6/609
Urinary tract infection (Infections and infestations) | 2/602 | 3/609
Animal bite (Injury, poisoning and procedural complications) | 1/602 | 0/609
Arthropod bite (Injury, poisoning and procedural complications) | 0/602 | 1/609
Fibula fracture (Injury, poisoning and procedural complications) | 0/602 | 1/609
Joint sprain (Injury, poisoning and procedural complications) | 1/602 | 0/609
Tooth fracture (Injury, poisoning and procedural complications) | 1/602 | 0/609
Blood pressure increased (Investigations) | 1/602 | 2/609
Gastric pH decreased (Investigations) | 0/602 | 1/609
Liver palpable subcostal (Investigations) | 1/602 | 0/609
Pulse abnormal (Investigations) | 0/602 | 1/609
Weight increased (Investigations) | 0/602 | 1/609
Gout (Metabolism and nutrition disorders) | 1/602 | 0/609
Hyperkalaemia (Metabolism and nutrition disorders) | 0/602 | 1/609
Hyponatraemia (Metabolism and nutrition disorders) | 0/602 | 1/609
Impaired fasting glucose (Metabolism and nutrition disorders) | 0/602 | 1/609
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 4/602 | 1/609
Arthralgia (Musculoskeletal and connective tissue disorders) | 2/602 | 3/609
Back pain (Musculoskeletal and connective tissue disorders) | 3/602 | 2/609
Bursitis (Musculoskeletal and connective tissue disorders) | 1/602 | 0/609
Joint contracture (Musculoskeletal and connective tissue disorders) | 0/602 | 1/609
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0/602 | 1/609
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3/602 | 0/609
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0/602 | 1/609
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1/602 | 0/609
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 3/602 | 0/609
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3/602 | 0/609
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1/602 | 0/609
Myalgia (Musculoskeletal and connective tissue disorders) | 6/602 | 12/609
Neck pain (Musculoskeletal and connective tissue disorders) | 2/602 | 0/609
Synovitis (Musculoskeletal and connective tissue disorders) | 0/602 | 1/609
Tendonitis (Musculoskeletal and connective tissue disorders) | 0/602 | 1/609
Torticollis (Musculoskeletal and connective tissue disorders) | 0/602 | 1/609
Balance disorder (Nervous system disorders) | 0/602 | 1/609
Burning sensation (Nervous system disorders) | 1/602 | 0/609
Carpal tunnel syndrome (Nervous system disorders) | 1/602 | 0/609
Dizziness (Nervous system disorders) | 9/602 | 7/609
Headache (Nervous system disorders) | 6/602 | 11/609
Hypoaesthesia (Nervous system disorders) | 2/602 | 1/609
Lethargy (Nervous system disorders) | 1/602 | 1/609
Loss of consciousness (Nervous system disorders) | 0/602 | 1/609
Paraesthesia (Nervous system disorders) | 12/602 | 2/609
Post herpetic neuralgia (Nervous system disorders) | 0/602 | 1/609
Sciatica (Nervous system disorders) | 2/602 | 1/609
Somnolence (Nervous system disorders) | 0/602 | 1/609
Syncope (Nervous system disorders) | 1/602 | 0/609
Tremor (Nervous system disorders) | 0/602 | 1/609
Anger (Psychiatric disorders) | 1/602 | 0/609
Anxiety (Psychiatric disorders) | 1/602 | 2/609
Depression (Psychiatric disorders) | 0/602 | 1/609
Insomnia (Psychiatric disorders) | 3/602 | 6/609
Dysuria (Renal and urinary disorders) | 1/602 | 0/609
Haematuria (Renal and urinary disorders) | 0/602 | 1/609
Nephrolithiasis (Renal and urinary disorders) | 1/602 | 1/609
Breast pain (Reproductive system and breast disorders) | 0/602 | 1/609
Menstruation delayed (Reproductive system and breast disorders) | 0/602 | 1/609
Asthma (Respiratory, thoracic and mediastinal disorders) | 1/602 | 0/609
Cough (Respiratory, thoracic and mediastinal disorders) | 3/602 | 2/609
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1/602 | 0/609
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2/602 | 1/609
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1/602 | 0/609
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0/602 | 1/609
Acne (Skin and subcutaneous tissue disorders) | 1/602 | 0/609
Acrodermatitis (Skin and subcutaneous tissue disorders) | 1/602 | 0/609
Alopecia (Skin and subcutaneous tissue disorders) | 1/602 | 0/609
Dandruff (Respiratory, thoracic and mediastinal disorders) | 0/602 | 1/609
Dermatitis (Skin and subcutaneous tissue disorders) | 2/602 | 0/609
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1/602 | 0/609
Drug eruption (Skin and subcutaneous tissue disorders) | 1/602 | 1/609
Eczema (Skin and subcutaneous tissue disorders) | 1/602 | 1/609
Erythema (Skin and subcutaneous tissue disorders) | 6/602 | 3/609
Heat rash (Skin and subcutaneous tissue disorders) | 0/602 | 1/609
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2/602 | 0/609
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1/602 | 0/609
Night sweats (Skin and subcutaneous tissue disorders) | 0/602 | 1/609
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1/602 | 0/609
Pruritus (Skin and subcutaneous tissue disorders) | 52/602 | 10/609
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2/602 | 0/609
Rash (Skin and subcutaneous tissue disorders) | 11/602 | 0/609
Rash erythematous (Skin and subcutaneous tissue disorders) | 1/602 | 2/609
Rash generalised (Skin and subcutaneous tissue disorders) | 1/602 | 0/609
Rash macular (Skin and subcutaneous tissue disorders) | 0/602 | 1/609
Rash pruritic (Skin and subcutaneous tissue disorders) | 0/602 | 1/609
Rosacea (Skin and subcutaneous tissue disorders) | 0/602 | 1/609
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0/602 | 1/609
Skin burning sensation (Skin and subcutaneous tissue disorders) | 3/602 | 0/609
Skin discolouration (Skin and subcutaneous tissue disorders) | 1/602 | 0/609
Skin irritation (Skin and subcutaneous tissue disorders) | 1/602 | 1/609
Swelling face (Surgical and medical procedures) | 1/602 | 0/609
Urticaria (Skin and subcutaneous tissue disorders) | 1/602 | 2/609
Blood pressure fluctuation (Vascular disorders) | 0/602 | 1/609
Flushing (Vascular disorders) | 68/602 | 9/609
Hypertension (Vascular disorders) | 0/602 | 1/609
Orthostatic hypotension (Vascular disorders) | 1/602 | 0/609
Phlebitis (Vascular disorders) | 0/602 | 1/609
Varicose vein (Vascular disorders) | 1/602 | 0/609
Alanine aminotransferase increased (Investigations) | 7/602 | 0/609
Aspartate aminotransferase increased (Investigations) | 5/602 | 1/609
Blood creatine phosphokinase increased (Investigations) | 4/602 | 0/609
Blood creatinine increased (Investigations) | 1/602 | 0/609
Blood glucose increased (Investigations) | 9/602 | 0/609
Blood lactate dehydrogenase increased (Investigations) | 1/602 | 0/609
Blood potassium increased (Investigations) | 0/602 | 1/609
Gamma-glutamyltransferase increased (Investigations) | 2/602 | 1/609

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.